CLINICAL TRIAL: NCT00313339
Title: AMORCYTE MYOCARDIAL REPAIR STUDY- A Phase I Trial of Intra-coronary Infusion of Bone Marrow Derived Autologous CD34+ Selected Cells in Patients With Acute Myocardial Infarction. (AMRS)
Brief Title: Intra-coronary Infusion of Bone Marrow Derived Autologous CD34+ Selected Cells in Patients With Acute Myocardial Infarction
Acronym: AMR-1
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Texas Heart Institute (Other)
Responsible Party: Principal Investigator, Arshed A. Quyyumi, Professor, Emory University
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 0076-2006; FDA IND 12584
Record Dates: First submitted 2006-04-10; First posted 2006-04-12 (Estimated); Last update posted 2013-11-18 (Estimated); Status verified 2013-11

CONDITIONS: Myocardial Infarction; Coronary Artery Disease
Keywords: myocardial infarction; bone marrow; cd34+; stem cells
MeSH Terms: conditions — Myocardial Infarction; Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control Group (No Intervention): A concurrent group meeting eligibility criteria but not receiving CD34+cells will be evaluated similar to the study group to assess the extent, if any, of significant improvement in cardiac perfusion/function without the CD34+cell product infusion.
- Treatment Group (Experimental): Intra-coronary infusion of an autologous bone marrow derived CD34+ stem cell product.
  Interventions: Drug: Intra-coronary infusion

INTERVENTIONS:
Drug: Intra-coronary infusion — In our study there will be four dosing cohorts (5, 10, 20 and 30 x 106) of CD34+ cells.
  Arms: Treatment Group

SUMMARY:
Following a Heart attack the acute loss of heart muscle cells results in a cascade of events causing an immediate decrease in cardiac function that has the potential to persist long term. Despite revascularization of the infarct related artery circulation and appropriate medical management to minimize the stresses on the heart walls, a significant percentage of patients experience permanent cardiac dysfunction and consequently remain at an increased life-time risk of experiencing adverse cardiac events, including death.

There is a great potential for stem cell therapy, using a variety of cell precursors (particularly hematopoietic,)to contribute to new blood vessel formation (and possibly limited heart muscle formation) and muscle preservation in the myocardial infarct zone. The administration of cells via an infusion through the infarct related artery appears to be feasible and result in a clinical effect in some studies.

Therefore, we propose to evaluate the safety and efficacy of a CD34+ selected stem cell product (AMR-001), administered through the infarct related coronary artery 6 to 9 days after successful infarct related artery stent placement.

The primary objective of the study is to determine the feasibility and safety of prospectively identifying patients at risk for clinically significant cardiac dysfunction following a myocardial infarction and the ability to isolate and infuse via the affected coronary circulation an autologous bone marrow derived CD34+ cell product at four dose levels.

The secondary objective of the study is to assess the effect on cardiac function and infarct region perfusion. A concurrent patient group meeting eligibility but not receiving CD34+ cells will be evaluated similar to the treated group to assess the rate of significant spontaneous improvement in cardiac function without CD34+cell infusion.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 - 75 years.
* Acute ST elevation myocardial infarction meeting ACC/AHA criteria, with symptoms of chest pain within 3 days of admission. Criteria include (ST elevation > 1mm in limb leads or 2 mm in two or more precordial leads and increased levels of troponin, CPK MB or both)
* NYHA heart failure class of I, II or III

Exclusion Criteria:

* Patients who are not candidates for percutaneous intervention, conscious sedation, MRI, SPECT imaging or mini-bone marrow harvest
* History of sustained chest pain unrelieved by nitrates, occurring 4 or more days before revascularization.
* Patients who fail to re-perfuse the infarct related coronary artery or have successful stent placement

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2006-03; Primary Completion 2009-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Cardiac function at 3 and 6 months follow-up will be compared to baseline measures obtained the day(s) before CD34+ cell product infusion. | 3 & 6 Months

SECONDARY OUTCOMES:
Perfusion of the infarct region at 6 months follow-up will be compared to baseline measures obtained the day(s) before CD34+ cell product infusion | 6 Months
An assessment will be performed to determine if a correlation exist between clinical outcome and cell content (CD34+) and/or in vitro colony growth (CFU-GM, CFU-GEMM, BFU-E) CXCR-4 mobility and CXCR-4 and/or VEGF surface antigen expression. | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: ARSHED A QUYYUMI, MD, Principal Investigator — Emory University
Locations (1):
- Emory University, Atlanta, Georgia, United States

REFERENCES:
- [Background] Quyyumi AA, Waller EK, Murrow J, Esteves F, Galt J, Oshinski J, Lerakis S, Sher S, Vaughan D, Perin E, Willerson J, Kereiakes D, Gersh BJ, Gregory D, Werner A, Moss T, Chan WS, Preti R, Pecora AL. CD34(+) cell infusion after ST elevation myocardial infarction is associated with improved perfusion and is dose dependent. Am Heart J. 2011 Jan;161(1):98-105. doi: 10.1016/j.ahj.2010.09.025. PMID 21167340
- [Result] Murrow J, Esteves F, Galt J, Chen J, Garcia E, Lin J, Lerakis S, Sher S, Khan Pohlel F, Waller EK, Vaughan D, Perin E, Willerson J, Kereiakes D, Preti R, Pecora AL, Quyyumi AA. Characterization of mechanical dyssynchrony measured by gated single photon emission computed tomography phase analysis after acute ST-elevation myocardial infarction. J Nucl Cardiol. 2011 Oct;18(5):912-9. doi: 10.1007/s12350-011-9414-8. Epub 2011 Jun 30. PMID 21717276